CLINICAL TRIAL: NCT02357901
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study To Assess the Efficacy, Safety, and Tolerability of Multiple Subcutaneous Injections of Depot Buprenorphine (RBP-6000 [100 mg and 300 mg]) Over 24 Weeks in Treatment-Seeking Subjects With Opioid Use Disorder
Brief Title: Treatment Seeking Participants With Opioid Use Disorders Assessing Tolerability of Depot Injections of Buprenorphine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RB-US-13-0001
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Results first posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Opioid Dependence; Opioid Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- RBP-6000 300mg/100mg (Experimental): During the Run-In Period, participants are inducted onto SUBOXONE sublingual film (SL) followed by a 4- to 11-day SUBOXONE sublingual film open-label run-in dose-adjustment period to achieve buprenorphine dosages ranging from 8 to 24 mg according to the SUBOXONE sublingual film prescribing information. Participants are then randomized. As of protocol Amendment 2 (21 August 2015) SUBOXONE use is tapered from 6 mg to 2 mg from Days 1-5 and then discontinued.
  Participants in this treatment arm are given RBP-6000 300 mg injections on Days 1 and 29. Injections 3-6 are separated by 28 days (Day 57-Day 141) and contain RBP-6000 100 mg.
  In addition, participants received individual drug counseling (IDC) at least once a week.
  Interventions: Drug: SUBOXONE; Drug: RBP-6000
- RBP-6000 300mg/300mg (Experimental): During the Run-In Period, participants are inducted onto SUBOXONE sublingual film (SL) followed by a 4- to 11-day SUBOXONE sublingual film open-label run-in dose-adjustment period to achieve buprenorphine dosages ranging from 8 to 24 mg according to the SUBOXONE sublingual film prescribing information. Participants are then randomized. As of protocol Amendment 2 (21 August 2015) SUBOXONE use is tapered from 6 mg to 2 mg from Days 1-5 and then discontinued.
  Participants in this treatment arm are given six RBP-6000 300 mg injections on Days 1 to 141 with injections separated by 28 days.
  In addition, participants received individual drug counseling (IDC) at least once a week.
  Interventions: Drug: SUBOXONE; Drug: RBP-6000
- Placebo Matching 300 mg/100 mg RBP-6000 (Placebo Comparator): During the Run-In Period, participants are inducted onto SUBOXONE sublingual film (SL) followed by a 4- to 11-day SUBOXONE sublingual film open-label run-in dose-adjustment period to achieve buprenorphine dosages ranging from 8 to 24 mg according to the SUBOXONE sublingual film prescribing information. Participants are then randomized. As of protocol Amendment 2 (21 August 2015) SUBOXONE use is tapered from 6 mg to 2 mg from Days 1-5 and then discontinued.
  Participants in this treatment arm are given placebo injections on Days 1 and 29 (matching the RBP-6000 300 mg dose volume). Injections 3-6 are separated by 28 days (Day 57-Day 141) and also contain placebo (matching the RBP-6000 100 mg volume).
  In addition, participants received individual drug counseling (IDC) at least once a week.
  Interventions: Drug: SUBOXONE; Drug: Placebo
- Placebo Matching 300 mg RBP-6000 (Placebo Comparator): During the Run-In Period, participants are inducted onto SUBOXONE sublingual film (SL) followed by a 4- to 11-day SUBOXONE sublingual film open-label run-in dose-adjustment period to achieve buprenorphine dosages ranging from 8 to 24 mg according to the SUBOXONE sublingual film prescribing information. Participants are then randomized. As of protocol Amendment 2 (21 August 2015) SUBOXONE use is tapered from 6 mg to 2 mg from Days 1-5 and then discontinued.
  Participants in this treatment arm are given six placebo injections (volume-matched to RBP-6000 300 mg dose) on Days 1 to 141 with injections separated by 28 days.
  In addition, participants received individual drug counseling (IDC) at least once a week.
  Interventions: Drug: SUBOXONE; Drug: Placebo

INTERVENTIONS:
Drug: SUBOXONE — SUBOXONE (buprenorphine sublingual film) is used for induction therapy. Participants take sublingual film for 3 days according to the sublingual film prescribing information; they then complete a 4-to-11 day sublingual film dose adjustment at doses ranging from 8 mg to 24 mg sublingual film prior to randomization. Following randomization, SUBOXONE use is tapered from 6 mg to 2 mg from Days 1-5 and then discontinued.
  Other Names: buprenorphine; Sublingual Film
Drug: RBP-6000 — Six injections administered subcutaneously every 28 days on alternate sides of participant's abdomen at either 300 mg or 100 mg dose.
  Other Names: Buprenorphine
  Arms: RBP-6000 300mg/100mg; RBP-6000 300mg/300mg
Drug: Placebo — Six injections of placebo administered subcutaneously every 28 days on alternate sides of participant's abdomen at volumes matching the experimental drug.
  Other Names: Volume-matched placebo
  Arms: Placebo Matching 300 mg RBP-6000; Placebo Matching 300 mg/100 mg RBP-6000

SUMMARY:
This is a randomized, double-blind, placebo controlled, multicenter study in male and female participants who are seeking treatment for opioid use disorder.

DETAILED DESCRIPTION:
After completing an up to 2-week screening period, subjects entered an open-label run-in induction phase with SUBOXONE (buprenorphine/naloxone) sublingual film for 3 days followed by a 4- to 11-day SUBOXONE sublingual film open-label run-in dose-adjustment period to achieve buprenorphine dosages ranging from 8 to 24 mg according to the SUBOXONE sublingual film prescribing information.

This is a 24-week non-residential study with participants being randomized after meeting randomization criteria. On Day 1 and Day 29 (± 2 days) participants will receive subcutaneous injections of 300 mg RBP-6000 or placebo. Thereafter, participants will receive 4 injections (once every 28 days ± 2 days) of either 300 mg or 100 mg RBP-6000 doses or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Currently meets Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for moderate or severe opioid use disorder
* By medical history has met DSM-5 criteria for moderate or severe opioid use disorder for the 3 months immediately prior to signing the informed consent form
* Is seeking medication-assisted treatment for opioid use disorder
* Is an appropriate candidate for opioid partial-agonist medication-assisted treatment in the opinion of the investigator or medically responsible physician
* Body mass index (BMI) of ≥ 18.0 to ≤ 35.0 kg/m^2

Exclusion Criteria:

* Current diagnosis other than opioid use disorder requiring chronic opioid treatment
* Current substance use disorder as defined by DSM-5 criteria with regard to any substances other than opioids, cocaine, cannabis, tobacco, or alcohol.
* Positive urine drug screen (UDS) result at screening for cocaine or cannabis AND meets DSM-5 criteria for either moderate or severe cocaine or cannabis use disorder, respectively
* Meets DSM-5 criteria for moderate or severe alcohol use disorder
* Received medication-assisted treatment for opioid use disorder (e.g., methadone, buprenorphine) in the 90 days prior to providing written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2016-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Global Clinical Development, Study Director — Indivior Inc.
Locations (38):
- United States (38):
  - Haleyville Clinical Research, Haleyville, Alabama
  - Boyett Health Services, Hamilton, Alabama
  - Woodland International Research Group, Little Rock, Arkansas
  - Collaborative Neuroscience Network, Garden Grove, California
  - Behavioral Research Specialists, Glendale, California
  - Synergy Clinical Research Center, National City, California
  - North County Clinical Research, Oceanside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Care Practice, San Francisco, California
  - Southern California Research, Thousand Oaks, California
  - Amit Vijapura, Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - Innovative Clinical Research, Lauderhill, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - Try Research, Maitland, Florida
  - Scientific Clinical Research, North Miami, Florida
  - Research Centers of America, Oakland Park, Florida
  - Behavioral Health Care Associates, Schaumburg, Illinois
  - Phoenix Medical Research, Prairie Village, Kansas
  - Louisiana Research Associates, New Orleans, Louisiana
  - Louisiana Clinical Research, Shreveport, Louisiana
  - Stanley Street Treatment and Resources, Fall River, Massachusetts
  - Adams Clinical Trials, Watertown, Massachusetts
  - Precise Research Centers, Inc., Flowood, Mississippi
  - St Louis Clinical Trials, St Louis, Missouri
  - Altea Research, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Neuro-behavioral Clinical Research, Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Charak Clinical Research Center, Garfield Heights, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Pahl Pharmaceutical Professionals, Oklahoma City, Oklahoma
  - CODA, Portland, Oregon
  - Tipton Medical and Diagnostic Center aka Clinical Research Associates of Central PA, Altoona, Pennsylvania
  - UPenn Treatment Research Center, Philadelphia, Pennsylvania
  - Carolina Clinical Trials, Charleston, South Carolina
  - Pillar Clinical Research, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greenwald MK, Wiest KL, Haight BR, Laffont CM, Zhao Y. Examining the benefit of a higher maintenance dose of extended-release buprenorphine in opioid-injecting participants treated for opioid use disorder. Harm Reduct J. 2023 Dec 2;20(1):173. doi: 10.1186/s12954-023-00906-7. PMID 38042801
- [Derived] Rutrick D, Learned SM, Boyett B, Hassman D, Shinde S, Zhao Y. 18-Month efficacy and safety analysis of monthly subcutaneous buprenorphine injection for opioid use disorder: Integrated analysis of phase 3 studies. J Subst Use Addict Treat. 2023 Nov;154:209155. doi: 10.1016/j.josat.2023.209155. Epub 2023 Aug 30. PMID 37657559
- [Derived] Laffont CM, Ngaimisi E, Gopalakrishnan M, Ivaturi V, Young M, Greenwald MK, Heidbreder C. Buprenorphine exposure levels to optimize treatment outcomes in opioid use disorder. Front Pharmacol. 2022 Nov 18;13:1052113. doi: 10.3389/fphar.2022.1052113. eCollection 2022. PMID 36467036
- [Derived] Craft WH, Tegge AN, Keith DR, Shin H, Williams J, Athamneh LN, Stein JS, Chilcoat HD, Le Moigne A, DeVeaugh-Geiss A, Bickel WK. Recovery from opioid use disorder: A 4-year post-clinical trial outcomes study. Drug Alcohol Depend. 2022 May 1;234:109389. doi: 10.1016/j.drugalcdep.2022.109389. Epub 2022 Mar 9. PMID 35287034
- [Derived] Boyett B, Wiest K, McLeod LD, Nelson LM, Bickel WK, Learned SM, Heidbreder C, Fudala PJ, Le Moigne A, Zhao Y. Assessment of craving in opioid use disorder: Psychometric evaluation and predictive validity of the opioid craving VAS. Drug Alcohol Depend. 2021 Dec 1;229(Pt B):109057. doi: 10.1016/j.drugalcdep.2021.109057. Epub 2021 Sep 24. PMID 34794061
- [Derived] Kranzler HR, Lynch KG, Crist RC, Hartwell E, Le Moigne A, Laffont CM, Andorn AC. A Delta-Opioid Receptor Gene Polymorphism Moderates the Therapeutic Response to Extended-Release Buprenorphine in Opioid Use Disorder. Int J Neuropsychopharmacol. 2021 Feb 15;24(2):89-96. doi: 10.1093/ijnp/pyaa069. PMID 32920647
- [Derived] Haight BR, Learned SM, Laffont CM, Fudala PJ, Zhao Y, Garofalo AS, Greenwald MK, Nadipelli VR, Ling W, Heidbreder C; RB-US-13-0001 Study Investigators. Efficacy and safety of a monthly buprenorphine depot injection for opioid use disorder: a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2019 Feb 23;393(10173):778-790. doi: 10.1016/S0140-6736(18)32259-1. Epub 2019 Feb 18. PMID 30792007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 36 sites in the United States screened subjects in this study. Three sites did not randomize any subjects.
  Analyses of RB-US-13-0001 were planned, conducted, and reported with pooled placebo groups.
Groups:
- Run-In Period: During the Run-In Period, participants were inducted onto SUBOXONE sublingual film followed by a 4- to 11-day SUBOXONE sublingual film open-label run-in dose-adjustment period to achieve buprenorphine dosages ranging from 8 to 24 mg according to the SUBOXONE sublingual film prescribing information.
- RBP-6000 300mg/100mg: Participants were given RBP-6000 300 mg injections on Days 1 and 29. Injections 3-6 were separated by 28 days (Day 57-Day 141) and contained RBP-6000 100 mg.
  As of protocol Amendment 2 (21 August 2015) SUBOXONE sublingual film use was tapered from 6 mg to 2 mg from Days 1-5 and then discontinued.
  In addition, participants received individual drug counseling (IDC) at least once a week.
- RBP-6000 300mg/300mg: Participants were given six RBP-6000 300 mg injections on Days 1 to 141 with injections separated by 28 days.
  As of protocol Amendment 2 (21 August 2015) SUBOXONE sublingual film use was tapered from 6 mg to 2 mg from Days 1-5 and then discontinued.
  In addition, participants received individual drug counseling (IDC) at least once a week.
- Combined Placebo: Participants randomized to either of the two placebo treatment arms were combined into this one treatment arm for reporting purposes. Analyses of 13-0001 were planned, conducted, and reported with pooled placebo groups. These participants were given six volume-matched placebo injections on Days 1 to 141 with injections separated by 28 days.
  As of protocol Amendment 2 (21 August 2015) SUBOXONE sublingual film use was tapered from 6 mg to 2 mg from Days 1-5 and then discontinued.
  In addition, participants received individual drug counseling (IDC) at least once a week.
Period: Run-In Period (Days -14 to Day -1)
Arm/Group | Run-In Period | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Started | 665 (Received at least one dose of SUBOXONE sublingual film.) | 0 | 0 | 0
Completed | 504 | 0 | 0 | 0
Not Completed | 161 | 0 | 0 | 0
Not completed — Run-In failures | 161 | 0 | 0 | 0
Period: Treatment Period (Day 1 to Week 24)
Arm/Group | Run-In Period | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Started | 0 | 203 | 201 | 100
Safety Analysis Set (Analyzed as treated.) | 0 | 203 | 201 | 100
Full Analysis Set (Analyzed as randomized. One site excluded from efficacy analyses due to compliance issues.) | 0 | 194 | 196 | 99
Completed | 0 | 125 | 129 | 34
Not Completed | 0 | 78 | 72 | 66
Not completed — Lost to Follow-up | 0 | 26 | 23 | 12
Not completed — Withdrawal by Subject | 0 | 20 | 21 | 18
Not completed — Lack of Efficacy | 0 | 3 | 5 | 18
Not completed — Adverse Event | 0 | 6 | 10 | 2
Not completed — Protocol Violation | 0 | 2 | 5 | 0
Not completed — Withdrawal symptoms | 0 | 1 | 1 | 3
Not completed — Non-compliance with study drug | 0 | 2 | 0 | 2
Not completed — Subject withdrawn by investigator | 0 | 1 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — site closed by sponsor, incarceration... | 0 | 17 | 6 | 7

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo | Total
Number analyzed (Participants) | 203 | 201 | 100 | 504
Age, Customized [Count of Participants; unit: Participants]
  >=18 to <30 years | 44 | 45 | 23 | 112
  >=30 to <45 years | 88 | 95 | 45 | 228
  >=45 to <60 years | 64 | 53 | 30 | 147
  >= 60 years | 7 | 8 | 2 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 66 | 35 | 168
  Male | 136 | 135 | 65 | 336
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 18 | 10 | 41
  Not Hispanic or Latino | 190 | 183 | 90 | 463
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 1 | 6
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 57 | 55 | 20 | 132
  White | 140 | 144 | 78 | 362
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Tobacco use [Count of Participants; unit: Participants]
  Yes | 187 | 186 | 93 | 466
  No | 16 | 15 | 7 | 38
Caffeine use [Count of Participants; unit: Participants]
  Yes | 187 | 185 | 95 | 467
  No | 16 | 16 | 5 | 37
Alcohol use [Count of Participants; unit: Participants]
  Yes | 160 | 160 | 81 | 401
  No | 43 | 41 | 19 | 103
Drug use history [Count of Participants; unit: Participants]
  Opioids | 203 | 201 | 100 | 504
  Cocaine | 94 | 80 | 42 | 216
  Amphetamines/ Methamphetamine | 53 | 29 | 19 | 101
  Methadone | 25 | 14 | 5 | 44
  Cannabinoids | 113 | 95 | 53 | 261
  Barbiturates | 3 | 1 | 0 | 4
  Buprenorphine | 20 | 16 | 6 | 42
  Benzodiazepines | 25 | 20 | 13 | 58
  Phencyclidine | 0 | 2 | 1 | 3
  Other | 2 | 6 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Distribution Function (CDF) of the Percentage of Urine Samples Negative for Opioids Combined With Self-Reports Negative for Illicit Opioid Use Collected From Week 5 Through Week 24
Description: Data represent the count of participants at various percentage abstinence levels. Abstinence was defined as urine samples being negative for opioids AND negative self-reports (obtained from Timeline Followback (TLFB) interviews) for illicit opioid use. The primary endpoint was based on visits in which paired urine samples and self-reports were expected for each subject as specified in the schedule of events. Missing urine drug screen(s) (UDS) samples and/or self-reports were considered as non-negative.
Time Frame: Weekly from Weeks 5-24
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 194 | 196 | 99
Participants
  >=0% | 194 | 196 | 99
  >=10% | 139 | 126 | 11
  >=20% | 115 | 111 | 7
  >=30% | 101 | 101 | 6
  >=40% | 90 | 90 | 6
  >=50% | 86 | 82 | 4
  >=60% | 78 | 70 | 4
  >=70% | 66 | 67 | 2
  >=80% | 55 | 57 | 2
  >=90% | 41 | 48 | 2
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test — significance at the 0.025 level
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test — significance at the 0.025 level

2. Secondary Outcome: Percentage of Participants Considered A Treatment Success
Description: Treatment success is defined as a participant having ≥80% of urine samples negative for opioids combined with self-reports negative for illicit opioid use between weeks 5-24.
Time Frame: Weeks 5-24
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 194 | 196 | 99
percentage of participants | 28.4 | 29.1 | 2.0
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Significance level of 0.05
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Significance level of 0.05

3. Secondary Outcome: Cumulative Distribution Function (CDF) of the Percentage of Urine Samples Negative for Opioids From Week 5 Through Week 24
Description: Data represent the count of participants at various percentage levels in which urine samples tested negative for opioids. All missing reports for urine samples were considered non-negative.
Time Frame: Weekly from Weeks 5-24
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 194 | 196 | 99
Participants
  >=0% | 194 | 196 | 99
  >=10% | 140 | 129 | 17
  >=20% | 120 | 114 | 9
  >=30% | 106 | 109 | 8
  >=40% | 97 | 98 | 7
  >=50% | 91 | 88 | 6
  >=60% | 82 | 74 | 5
  >=70% | 73 | 69 | 4
  >=80% | 64 | 61 | 4
  >=90% | 47 | 51 | 2
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test — Significance level of 0.05
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test — Significance level of 0.05

4. Secondary Outcome: Cumulative Distribution Function (CDF) of the Percentage of Self-Reports Negative for Illicit Opioid Use From Week 5 Through Week 24
Description: Data represent the count of participants at various percentage levels in which self-reports were negative for illicit use of opioids. Self-reports were obtained from Timeline Followback (TLFB) interviews. All missing self-reports were considered non-negative.
Time Frame: Weekly from Weeks 5-24
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 194 | 196 | 99
Participants
  >=0% | 194 | 196 | 99
  >=10% | 163 | 162 | 37
  >=20% | 155 | 152 | 29
  >=30% | 139 | 139 | 24
  >=40% | 132 | 132 | 20
  >=50% | 125 | 125 | 18
  >=60% | 120 | 117 | 17
  >=70% | 108 | 112 | 14
  >=80% | 102 | 101 | 9
  >=90% | 92 | 91 | 7
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test — Significance level of 0.05
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test — Significance level of 0.05

5. Secondary Outcome: Change From Baseline in the Opioid Craving Visual Analog Scale (VAS) Prior to Injections From Week 5 Through Week 24 Analyzed by Mixed Model for Repeated Measures
Description: The opioid craving scale was a 100 mm scale with 0= 'no craving' on the left end and 100= 'strongest craving ever' on the right end of the scale. Participants marked where along the scale reflected their craving for opioids. The full range of the change from baseline scale was therefore 100 (no craving at baseline, strongest craving during study) to -100 (strongest craving at baseline, no craving during study).
  Baseline was defined as the last non-missing value prior to subcutaneous injection on Day 1. The opioid craving VAS was completed each week; measurements were taken prior to dosing on weeks 5, 9, 13, 17 and 21.
  Negative change from baseline values indicate a lessening of craving symptoms.
  Change from baseline was analyzed using a mixed model for repeated measures (MMRM) with terms for treatment, visit, and treatment-by-visit interaction as factors and baseline value as a covariate. Center was included in the model as a random effect.
Time Frame: Baseline: Day 1 (prior to dosing), Weeks 5-24
Population: Full analysis set of participants who had available data on baseline score and change from baseline in any visit through week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 192 | 193 | 96
units on a scale | 2.1 (1.63) | -0.9 (1.63) | 11.5 (2.48)
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; Change from baseline was analyzed using a mixed model for repeated measures (MMRM) with terms for treatment, visit, and treatment-by-visit interaction as factors and baseline value as a covariate. Center was included in the model as a random effect; Test type: Superiority; p = 0.0003, mixed model for repeated measures — Significance level of 0.05; LSM difference = -9.4, 95% CI 2-sided [-14.56 to -4.30], Standard Error of Mean 2.62
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, mixed model for repeated measures — Significance level of 0.05; LSM difference = -12.4, 95% CI 2-sided [-17.51 to -7.28], Standard Error of Mean 2.61

6. Secondary Outcome: Participants Who Complete the Week 24 Visit ("Completers")
Description: A completer was defined as a participant who completed either the urine drug screen (UDS) or Timeline Followback (TLFB) assessment at the Week 24 visit.
Time Frame: Week 24
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 194 | 196 | 99
Participants | 119 | 126 | 33
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; stratified by site
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; stratified by site

7. Secondary Outcome: Participants Who Are Abstinent at Week 24
Description: Participants with both a negative urine sample and negative self-report for illicit opioid use at Week 24.
Time Frame: Week 24
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 194 | 196 | 99
Participants | 71 | 87 | 2
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; stratified by site
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; stratified by site

8. Secondary Outcome: Change From Baseline in the Clinical Global Impression - Improvement Scale (CGI-I) Prior to Injections From Week 5 Through Week 24 Analyzed by Mixed Model for Repeated Measures
Description: The CGI-I was used to rate the change in clinical status since the start of the treatment on an ordinal scale ranging from 1 (very much improved; nearly all better; good level of functioning; minimal symptoms; represents a very substantial change) to 7 (very much worse; severe exacerbation of symptoms and loss of functioning). Baseline was defined as the last non-missing value prior to subcutaneous injection on Day 1. Measurements taken during the treatment period were taken at the end of each 28 day treatment and prior to dosing of the next treatment.
  Negative change from baseline values indicate an improved clinical global impression.
  Change from baseline was analyzed using a mixed model for repeated measures (MMRM) with terms for treatment, visit, and treatment-by-visit interaction as factors and baseline value as a covariate. Center was included in the model as a random effect.
Time Frame: Baseline: Day 1 (prior to dosing), Days 29, 57, 85, 113, 141, 169
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 169 | 173 | 60
units on a scale | 1.6 (0.11) | 1.5 (0.11) | 2.4 (0.15)
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.7, 95% CI 2-sided [-0.96 to -0.46], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.9, 95% CI 2-sided [-1.12 to -0.62], Standard Error of Mean 0.13

9. Secondary Outcome: Change From Baseline in the Clinical Global Impression - Severity Scale (CGI-S) Prior to Injections From Week 5 Through Week 24 Analyzed by Mixed Model for Repeated Measures
Description: The CGI-S was an assessment completed by the clinician to rate the severity of symptoms on an ordinal scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill subjects; pathology drastically interferes in many life functions). Baseline was defined as the last non-missing value prior to subcutaneous injection on Day 1. Measurements taken during the treatment period were taken at the end of each 28 day treatment and prior to dosing of the next treatment.
  Negative change from baseline values indicate an improvement in the severity of symptoms.
  Change from baseline was analyzed using a mixed model for repeated measures (MMRM) with terms for treatment, visit, and treatment-by-visit interaction as factors and baseline value as a covariate. Center was included in the model as a random effect.
Time Frame: Baseline: Day 1 (prior to dosing), Days 29, 57, 85, 113, 141, 169
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 166 | 170 | 59
units on a scale | -0.7 (0.13) | -0.7 (0.13) | -0.0 (0.17)
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.6, 95% CI 2-sided [-0.89 to -0.33], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.7, 95% CI 2-sided [-0.97 to -0.41], Standard Error of Mean 0.14

10. Secondary Outcome: Change From Baseline in the Clinical Opiate Withdrawal Scale (COWS) Through Week 24 Analyzed by Mixed Model for Repeated Measures
Description: COWS is an 11-item instrument used to assess signs and symptoms of opioid withdrawal (Wesson et al., 1999). The score is the sum of the responses for a total range of 0-48. The COWS is commonly used by clinicians treating patients with buprenorphine to monitor the severity of withdrawal. COWS scores below 5 are considered not indicative of withdrawal. Scores from 5 to 12 are considered mild withdrawal; from 13 to 24 moderate withdrawal; 25 to 36 moderately severe withdrawal, and 37-48 severe withdrawal. Negative change from baseline values indicate a lessening of withdrawal symptoms.
  Baseline was defined as the last non-missing value prior to subcutaneous injection on Day 1. The COWS was completed each week; measurements were taken prior to dosing on weeks 5, 9, 13, 17 and 21.
  Change from baseline was analyzed using a mixed model for repeated measures (MMRM) with terms for treatment, visit, and treatment-by-visit interaction as factors and baseline value as a covariate.
Time Frame: Baseline: Day 1 (prior to dosing), Baseline: Day 1 (prior to dosing), Days 2, 8, 5, 22, 29, 30, 36, 43, 50, 57, 58, 64, 71, 78, 85, 86, 92, 99, 106, 113, 114, 120, 127, 134, 141, 142, 148, 155, 162, 169
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 191 | 192 | 96
units on a scale | -0.5 (0.22) | -1.1 (0.21) | -0.1 (0.35)
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.3143, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.4, 95% CI 2-sided [-1.13 to 0.36], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0101, mixed model for repeated measures — Significance level of 0.05; LSM difference = -1.0, 95% CI 2-sided [-1.72 to -0.23], Standard Error of Mean 0.38

11. Secondary Outcome: Change From Baseline in the Subjective Opiate Withdrawal Scale (SOWS) Through Week 24 Analyzed by Mixed Model for Repeated Measures
Description: The Subjective Opiate Withdrawal Scale (SOWS) contains 16 symptoms whose intensity the participant rates on a scale of 0 (not at all) to 4 (extremely) for a full scale of 0 (no withdrawal symptoms) to 64 (extreme withdrawal symptoms). Negative change from baseline values indicate a lessening of withdrawal symptoms.
  Baseline was defined as the last non-missing value prior to subcutaneous injection on Day 1. The SOWS was completed each week; measurements were taken prior to dosing on weeks 5, 9, 13, 17 and 21.
  Change from baseline was analyzed using a mixed model for repeated measures (MMRM) with terms for treatment, visit, and treatment-by-visit interaction as factors and baseline value as a covariate.
Time Frame: as for outcome 10
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 192 | 193 | 96
units on a scale | -0.9 (0.51) | -2.0 (0.51) | 0.7 (0.80)
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0726, mixed model for repeated measures — Significance level of 0.05; LSM difference = -1.6, 95% CI 2-sided [-3.29 to 0.14], Standard Error of Mean 0.87
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0028, mixed model for repeated measures — Significance level of 0.05; LSM difference = -2.6, 95% CI 2-sided [-4.32 to -0.90], Standard Error of Mean 0.87

12. Secondary Outcome: Total Number of Weeks of Abstinence as Assessed From Urine Samples Negative for Opioids Combined With Self-Reports Negative for Illicit Opioid Use Collected From Week 5 Through Week 24
Description: The total number of weeks of abstinence was assessed from urine samples negative for opioids combined with self-reports negative for illicit opioid use collected from week 5 through week 24. All missing reports for opioids were considered non-negative.
Time Frame: Weeks 5 through 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: weeks
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 194 | 196 | 99
weeks | 8.5 (0.68) | 8.5 (0.68) | 1.0 (0.84)
Statistical Analysis 1: Comparison: RBP-6000 300mg/100mg vs Combined Placebo; Test type: Superiority; p < 0.0001, ANOVA — Significance level of 0.05; a random effects ANOVA model with treatment included as fixed effect and center as random effect; LSM difference = 7.5, 95% CI 2-sided [5.81 to 9.20], Standard Error of Mean 0.86
Statistical Analysis 2: Comparison: RBP-6000 300mg/300mg vs Combined Placebo; Test type: Superiority; p < 0.0001, ANOVA — Significance level of 0.05; a random effects ANOVA model with treatment included as fixed effect and center as random effect; LSM difference = 7.5, 95% CI 2-sided [5.82 to 9.21], Standard Error of Mean 0.86

13. Secondary Outcome: Participants With Adverse Events During the Treatment Period
Description: Treatment-emergent adverse event (TEAE) = any untoward medical occurrence that develops or worsens in severity after dispensation of the study drug and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= a marked limitation in activity. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 1 through Week 24
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 203 | 201 | 100
Participants
  >=1 TEAE | 155 | 134 | 56
  >=1 TEAE related to study drug | 67 | 70 | 23
  >=1 serious TEAE | 4 | 7 | 5
  >=1 serious study treatment-related TEAE | 0 | 0 | 0
  Death | 0 | 1 | 0
  >=1 severe TEAE | 15 | 13 | 4
  TEAE leading to study treatment discontinuation | 7 | 10 | 2

14. Secondary Outcome: Worst Injection Site Pain From Injections 1-6 as Measured by Participant-Reported Visual Analog Scale (VAS)
Description: Injection site pain as measured by participant-reported VAS The participant-reported VAS for injection site pain was measured on a 100 mm scale with 'no pain' on the left end and 'strongest pain ever' on the right end of the scale (total scale of 0-100). Participants marked where along the scale reflected their localized injection pain.
  The injection site pain VAS scores were obtained (after the completion of the injection) within 1 minute and at 5, 10, 15, 30, 60 and 120 minutes (+- 5 minutes). The timing of the injection site pain VAS should have been measured from the end of the injection.
  Data represents the worst pain recorded for each participant across all 6 injections and all VAS records. The mean value is presented.
Time Frame: Days 1, 29, 57, 85, 113, 141
Population: Safety population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 202 | 201 | 100
units on a scale | 55.8 (27.07) | 63.3 (29.33) | 61.0 (28.79)

15. Secondary Outcome: Suicidality Using the Columbia Suicide Severity Rating Scale (C-SSRS) From Week 2 - 24
Description: The C-SSRS asks questions of study participants regarding whether they had suicidal ideation and/or suicidal behavior since the last visit using the electronic version of the scale. The C-SSRS was completed each week; measurements were taken prior to dosing on weeks 5, 9, 13, 17 and 21.
Time Frame: Weekly - Week 2 through Week 24
Population: Safety analysis set of participants who completed a C-SSRS during the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
Number analyzed (Participants) | 202 | 200 | 98
Participants
  Suicidal Ideation: Wish to be dead | 15 | 11 | 9
  Non-specific active suicidal thoughts | 6 | 1 | 2
  (subset of above) No plan nor intent to act: number analyzed (Participants) | 6 | 1 | 2
  (subset of above) No plan nor intent to act | 2 | 0 | 1
  (subset of above) Non-specific plan, some intent: number analyzed (Participants) | 6 | 1 | 2
  (subset of above) Non-specific plan, some intent | 3 | 0 | 1
  (subset of above) Specific plan and intent: number analyzed (Participants) | 6 | 1 | 2
  (subset of above) Specific plan and intent | 0 | 0 | 0
  Suicidal Behaviour: Preparatory acts or behaviour | 0 | 0 | 0
  Aborted attempt | 1 | 1 | 1
  Interrupted attempt | 1 | 1 | 1
  Actual attempt | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Week 24
Arm/Group | RBP-6000 300mg/100mg | RBP-6000 300mg/300mg | Combined Placebo
All-Cause Mortality (participants affected / at risk) | 0/203 | 1/201 | 0/100
Serious Adverse Events (participants affected / at risk) | 4/203 | 7/201 | 5/100
Other Adverse Events (participants affected / at risk) | 97/203 | 84/201 | 27/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RBP-6000 300mg/100mg (N=203) | RBP-6000 300mg/300mg (N=201) | Combined Placebo (N=100)
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1
Hernia (General disorders) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelomalacia (Nervous system disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RBP-6000 300mg/100mg (N=203) | RBP-6000 300mg/300mg (N=201) | Combined Placebo (N=100)
Headache (Nervous system disorders) | 19 | 17 | 6
Constipation (Gastrointestinal disorders) | 19 | 16 | 0
Nausea (Gastrointestinal disorders) | 18 | 16 | 5
Injection site pruritus (General disorders) | 13 | 19 | 4
Vomiting (Gastrointestinal disorders) | 19 | 11 | 4
Insomnia (Psychiatric disorders) | 13 | 17 | 11
Upper respiratory tract infection (Infections and infestations) | 15 | 12 | 1
Injection site pain (General disorders) | 10 | 12 | 3
Nasopharyngitis (Infections and infestations) | 11 | 10 | 1
Fatigue (General disorders) | 8 | 12 | 3
Blood creatine phosphokinase increased (Investigations) | 11 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multi-center publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.